CLINICAL TRIAL: NCT04769947
Title: Observational Study in Adult Patient With Chronic Myeloid Leukemia Who Discontinue Tyrosine Kinase Inhibitors in Italy
Brief Title: Italian Treatment Free Remission Registry
Status: Recruiting | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: ITALY-TFR
Record Dates: First submitted 2021-02-10; First posted 2021-02-25 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-05

CONDITIONS: Treatment Free Remission; Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Cohort 1 retrospective/prospective study: 293 patients enrolled and reported in Fava et al 2019 (1) with at least 1 year of follow up at the end of the study (February 2017) and 107 patients enrolled but not reported in Fava et al 2019 since their follow-up was shorter than 1 year. The data for these patients will be collected since the end of previous study.
- Cohort 2: Cohort 2 retrospective/prospective study: patient not enrolled in the previous study (Fava et al 2019). The data for these patients will be collected since patient diagnosis to the end of the study.
- Cohort 3: Cohort 3 prospective study: patients who have discontinued TKI therapy after the study approval in each center. These patients will also participate in the validation process of Phase 2 of a questionnaire developed by an expert panel of eight CML patients with the purpose of capturing the experiences of people along all phases of the TFR.

SUMMARY:
The investigator propose an extension of the previous National, multicentric study, promoting an observational registry, both retrospective and prospective, in order to expand and further characterize the series of Italian patients with Philadelphia-positive, chronic phase CML (CP-CML) who discontinue TKIs in an off-protocol setting. As safety concerns may arise for patients receiving long-term treatments, and due to the growing number of patients discontinuing TKIs in clinical practice, the study aim to collect all available data regarding feasibility and freedom from progression of the cohort of patients.

DETAILED DESCRIPTION:
This is an observational, retrospective and prospective study of CP-CML patients who discontinue TKIs in Italy. The study will not imply additional costs for the participating centers. Data already present in the clinical charts will be collected.

The patients, answering to inclusion/exclusion criteria will be enrolled in one of the follow cohorts

* Cohort 1 retrospective/prospective study: 293 patients enrolled and reported in Fava et al 2019 with at least 1 year of follow up at the end of the study (February 2017) and 107 patients enrolled but not reported in Fava et al 2019 since their follow-up was shorter than 1 year. The data for these patients will be collected since the end of previous study.
* Cohort 2 retrospective/prospective study: patient not enrolled in the previous study (Fava et al 2019). The data for these patients will be collected since patient diagnosis to the end of the study.
* Cohort 3 prospective study: patients who have discontinued TKI therapy after the study approval in each center. These patients will also participate in the validation process of Phase 2 of a questionnaire developed by an expert panel of eight CML patients with the purpose of capturing the experiences of people along all phases of the TFR.

Patients participating in the study will not be subjected to any procedure that falls outside the clinical practice; in the same way, clinical variables that will be collected for the study are those that are commonly collected by physician in daily clinical practice.

Any decision about drug administration or suspension is made by the physician based on his clinical judgment in the context of clinical practice, independently from decision to include the patient in this study.

Registration of enrolled patients will be done on-line on a key restricted accessible web-database.

Primary objective and endpoint To assess the TFR rate at 1 year from discontinuation of TKIs. Secondary objectives and endpoints

* To further describe the observed population of patients in terms of:

  * treatment-free duration; o survival in MR4.5;
  * survival in MR3;
  * event-free survival;
  * progression-free survival;
  * deaths after treatment discontinuation;
  * rate of achievement of MMR and DMR after treatment re-initiation
* To identify clinical and biological prognostic factors affecting the persistence of off-therapy remission.
* To identify optimal timing and modalities of molecular monitoring of BCR-ABL1 transcript

  * Evaluation of the safe minimum monitoring during and after treatment discontinuation
  * Evaluation of the maximum MRD positivity level acceptable to safely stay off-treatment
* Evaluation of short-term adverse events (withdrawal syndrome: fever, arthralgia, myalgia, bone pain, weight loss) after treatment discontinuation
* Evaluation of long-term adverse events (i.e. cardiovascular adverse events, second neoplasia) after treatment discontinuation
* Validation of the Italian version of the "Phase 2" of a questionnaire developed by an expert panel of eight CML patients to capture the experiences of people along all phases of the TFR
* Evaluation of patient-reported outcomes describing quality of life of patients off therapy and after resumption of TKIs

ELIGIBILITY:
Inclusion Criteria:

* Patients with CP-CML, treated with TKI monotherapy or TKI in association with other drugs (such as interferon, BCR-ABL1 peptidic vaccine and others)
* Treatment with TKI discontinued for any reason
* Deep Molecular Response (DMR), defined as MR4 (BCR-ABL1 ratio ≤ 0.01% with at least 10,000 ABL1 copies), or MR4.5 (BCR-ABL1 ratio ≤ 0.0032% with at least 32,000 ABL1 copies), or MR5 (BCR-ABL1 ratio ≤ 0.001% with at least 100,000 ABL1 copies), confirmed at least three times before TKI discontinuation. In patients who discontinued TKIs before the establishment of molecular standardization, DMR will be defined as a level of BCR-ABL1 transcript undetectable by qPCR or by qualitative PCR, confirmed in at least two controls.
* Participant is willing and able to give informed consent for participation in the study Data regarding patients discontinuing in less than DMR (as defined above) will be collected and analysed separately.

Exclusion Criteria:

* Patients who were diagnosed with accelerated or blastic phase CML will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with CP-CML who discontinued treatment with TKIs in Italy will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-07-08 (Estimated); Study Completion 2030-02-08 (Estimated)

PRIMARY OUTCOMES:
TFR rate at 1 year from discontinuation of TKIs | 1 year
  To assess the TFR rate at 1 year from discontinuation of TKIs

SECONDARY OUTCOMES:
Secondary objectives | 10 years
  treatment-free duration (months); survival in MR4.5 (%); survival in MR3 (%); event-free survival (%); progression-free survival (%); deaths after treatment discontinuation (%); rate of achievement of MMR and DMR after treatment re-initiation (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Hematology-AO Mauriziano Hospital, University of Turin, Turin, Italy